CLINICAL TRIAL: NCT01406496
Title: The Effect of Food Content and Optimal Timing of Pre-meal Insulin Bolus on the Postprandial Glycemic Control in Children With Type 1 Diabetes
Brief Title: Best Timing of Insulin Bolus Before Meals of Different Contents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Amnon Zung, MD, Kaplan Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PP1
Record Dates: First submitted 2011-06-16; First posted 2011-08-01 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin bolus; glucose excursions; post-prandial; timing; meal content
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Timing of insulin administration (Experimental)
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: insulin — Three different timings of insulin delivered by a pump
  Other Names: Insulin Humalog (generic name Lispro); By Elli Lilly, USA

SUMMARY:
Post-meal glucose excursions may contribute to the development of diabetes-related complications. These glucose excursions are affected by the food content of the meal and the timing of insulin injection (or insulin pump-bolus) before meal. The best timing for insulin bolus (by pump) is controversial.

The aim of the study is to examine three different timings of insulin bolus in three types of breakfast meals that contain carbohydrates, carbohydrates + proteins and carbohydrate+ fat. The 3h post-meal glucose excursions will be recorded by continuous glucose monitoring system. The results obtained in the diabetic patients will be compared to those obtained in a group of healthy individuals that will consume similar meals.

ELIGIBILITY:
Inclusion Criteria:

Diabetes patients:

* Type 1 diabetes
* Age 8 to 20 years
* Both genders

Control group:

* Age 18 to 30 years
* Both genders

Exclusion Criteria:

Diabetes patients:

* Less than a year from the diagnosis of type 1 diabetes
* Less than 6 months from the time of insulin pump introduction

Control group:

* Pregnancy
* Any diagnosed or suspected chronic diseases
* Current or recent (within 1 month) use of drugs (not including oral contraceptives and inhaled steroids for asthma).

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Post-prandial blood glucose excursions following three different meals and three different timings of insulin bolus. | outcome measures will be assessed for each particiapant after a week; the overall timeframe for all participants is 18 months
  Each diabetes patient will be assigned for one of three breakfast meals, differed by their content: carbohydrates, carbohydrates + proteins or carbohydrates + fat. Post-meal blood glucose excursions will be recoded by continuous blood glucose monitoring at three different days. In each day insulin bolus will be administrated at a different timing before meal.
  Each healthy participant will consume the three types of breakfast meals at three different days, and post-meal blood glucose excursions will be recoded by continuous blood glucose monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Zung, MD, Principal Investigator — Pediatric Endocrinology Unit, Kaplan Medical Center, affiliated with the Hebrew University of Jerusalem
Locations (1):
- Pediatric Endocrinology Unit, Kaplan Medical Center, Rehovot, Israel